CLINICAL TRIAL: NCT03684291
Title: Effects of Two Different Ventilation Modes Used in Gynecologic Laparoscopic Operations Performed in Steep Trendelenburg Position on Hemodynamic Parameters
Brief Title: Hemodynamic Effects of Ventilation Modes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Hakan Yılmaz, Associate Professor, Ufuk University
Other Study IDs: HemodynamicsTrendelenburg
Record Dates: First submitted 2018-01-15; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Respiration, Artificial; Laparoscopy; Hemodynamics
Keywords: Mechanical ventilation; Laparoscopic surgery; Hemodynamics
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group V: The patients in this group are ventilated using VCV (Volume Control Ventilation) mode (FiO2 50%, Tidal volume: 6-8 ml/kg (ideal body weight), frequency: 12/minute, I/E ratio: 1/2, PEEP not applied)
  Interventions: Procedure: Mode of Mechanical Ventilation
- Group P: The patients in this group are ventilated using PCV-VG (Volume Guaranteed Pressure Control Ventilation) mode (FiO2 50%, Tidal volume: 6-8 ml/kg (ideal body weight), frequency: 12/minute (EtCO2 kept between 35-40 mmHg), Pressure limit: 30 cm H2O, I/E:1/2, PEEP not applied)
  Interventions: Procedure: Mode of Mechanical Ventilation

INTERVENTIONS:
Procedure: Mode of Mechanical Ventilation — Adjustment of mechanical ventilation mode

SUMMARY:
Different ventilation modes can be used in laparoscopic surgeries. These surgeries are performed in steep Trendelenburg position with serious hemodynamic disturbances. This study aims to observe the hemodynamic effects of two different ventilation modes in laparoscopic gynecologic surgery performed in steep Trendelenburg position.

ELIGIBILITY:
Inclusion Criteria:

* Women of ASA I and II classification between 18-65 years scheduled for elective gynecologic laparoscopic surgery

Exclusion Criteria:

* Patient refusal to participate
* Patients with severe cardiac (congestive heart failure etc) and pulmonary (COPD, pulmonary hypertension) disease (ASA > III)
* Morbid obesity
* Negative Allen test

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Observations will be performed in laparoscopic gynecological operations
Study Population: Women between 18 and 65 years of age scheduled to undergo elective gynecologic laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of changes in MAP | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Mean arterial pressure (MAP) (mmHg)
Measurement of changes in heart rate | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Heart rate (bpm)
Measurement of changes in systemic vascular resistance index | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Systemic vascular resistance index (dyne x sec/cm2)
Measurement of changes in stroke volume index | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Stroke volume index (mL/m2)
Measurement of changes in cardiac index | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Cardiac index L(min x m2)
Measurement of changes in stroke volume variation | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Stroke volume variation (%)
Measurement of changes in cardiac cycle efficiency | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Cardiac cycle efficiency (units)
Measurement of changes in aortic dp/dt | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Aortic dP/dt (mmHg/msec)

SECONDARY OUTCOMES:
Measurement of changes in peak airway pressure | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Ppeak (Peak airway pressure)
Measurement of changes in mean airway pressure | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Pmean (Mean Airway Pressure),
Measurement of changes in plateau airway pressure | T0: Induction (Baseline) T1: Change after 30 minutes pneumoperitoneum T2: Change after desufflation
  Pplateau (Plateau Airway Pressure)

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University Faculty of Medicine, Ankara, Balgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balderi T, Forfori F, Marra V, Di Salvo C, Dorigo M, Anselmino M, Romano SM, Giunta F. Continuous hemodynamic monitoring during laparoscopic gastric bypass in superobese patients by pressure recording analytical method. Obes Surg. 2008 Aug;18(8):1007-14. doi: 10.1007/s11695-007-9379-5. Epub 2008 Apr 15. PMID 18414959
- [Background] Liao CC, Kau YC, Ting PC, Tsai SC, Wang CJ. The Effects of Volume-Controlled and Pressure-Controlled Ventilation on Lung Mechanics, Oxidative Stress, and Recovery in Gynecologic Laparoscopic Surgery. J Minim Invasive Gynecol. 2016 Mar-Apr;23(3):410-7. doi: 10.1016/j.jmig.2015.12.015. Epub 2016 Jan 7. PMID 26772778